CLINICAL TRIAL: NCT05551234
Title: Reciprocal Benefit by Intergenerational Meetings Between 2 Fragile Populations
Brief Title: Reciprocal Benefit by Intergenerational Meetings
Acronym: Part'Ages
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 22CMRR01
Record Dates: First submitted 2022-09-09; First posted 2022-09-22 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Isolation, Social
MeSH Terms: conditions — Social Isolation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Isolated senior
  Interventions: Other: Regular exchanges
- Children
  Interventions: Other: Regular exchanges

INTERVENTIONS:
Other: Regular exchanges — The seniors and childrens will meet once a week, for 7 months, over a period of one and a half hours, outside school hours (4:30 p.m. to 6:00 p.m.) and school holidays.

SUMMARY:
The investigators want to set up an experiment that allows a reciprocal benefit to 2 fragile populations: isolated seniors and disadvantaged children. The main hypothesis is that regular exchanges between these two populations reduce the feeling of social isolation of seniors and improve the school behavior of childrens. Therefore the investigators propose the following study design. The seniors and childrens will meet once a week, for 7 months, in a defined location in the city of Vallauris, over a period of one and a half hours, outside school hours (4:30 p.m. to 6:00 p.m.) and school holidays. During the school holidays the group will meet 3 times for day-long activities in the presence of at least one of the parents and possibly brothers and sisters. At the end of the project, a convivial evening will be organized in the presence of the families. The group will meet in a room in the city center and in the presence of a facilitator so that an adult will never be alone with a child. The formed pair will follow a defined schedule where will alternate activities proposed by the senior, sessions proposed by the facilitator and convivial moments in the presence of families . During the sessions proposed by the senior, he will offered the child a leisure activity that he likes and masters (eg gardening, DIY, sewing, etc.). All the proposed activities will be validated upstream by the project managers. The sessions proposed by the facilitator (e.g. games, walks) could be done with the participation of an outside speaker (e.g. for writing a gazette). A new evaluation session will be offered to all participants at the end of the meeting period, then at the end of the project, 1 month after the end of the meeting period.

ELIGIBILITY:
Inclusion Criteria for children :

* Girls or boys from last year of kindergarten to last year of elementary school,
* Educated in priority education network,
* Having the cognitive and sensory-motor capacities to follow and interact during the workshops,

Exclusion Criteria for children :

- subject does not speak French, does not read French,

Inclusion Criteria for seniors:

* Men or women over the age of 65, - MMSE score greater than or equal to 24/30,
* A score above 4 on the 3-point Loneliness Scale (Three-item Loneliness Scale),
* Clean record.

Exclusion Criteria for Seniors:

* subject does not speak French, does not read French,
* subject with visual impairment,
* subject under guardianship or curatorship,

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: isolated seniors (from 65 years old) and disadvantaged children (from 5 years old)
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
For Senior : the 3-point loneliness scale; | At 8 months
  The 3-point lonelisness scale evaluates loneless with 3 questions.
For children : SDQ-fra | At 8 months
  The SDQ is a behavioral screening questionnaire applicable to children aged 3 to 16 and comprising 25 questions divided into 5 domains (emotional symptoms, conduct problems, hyperactivity/inattention, relationship problems with other children, social behavior).

SECONDARY OUTCOMES:
For Senior : the Nottingham Perceptual Health Indicator score (ISPN or NHP) | Before (Month 0), after the sessions (Month 7), one month after the end of the sessions (M8)
  This is a self-questionnaire of 38 items covering 6 dimensions: pain, physical mobility, sleep, energy, emotional reaction, social isolation. We will focus on the average score (and not the classes/slices: low, medium, etc.).
  This is a self-questionnaire of 38 items covering 6 dimensions: pain, physical mobility, sleep, energy, emotional reaction, social isolation. We will focus on the average score (and not the classes/slices: low, medium, etc.).
Geriatric depression scale 15 | Up to 8 months
  The GDS is a 15-item scale used to screen for mood disorders.
rosenberg self-esteem scale | Up to 8 months
  This scale consists of 10 questions each evaluated by a 4-level Likert scale.
satisfaction questionnaire | At 7 months
  for children and their parents and teachers, for the senior
semi-directive interiew | Up to 7 months
  "for children, for the senior, for entourage of senior and children interview defined especially for this study to evaluate social impact written transcription or oral records"

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Claude Pompidou, Nice, France

IPD SHARING:
Plan to Share IPD: No
IPD sharing is not planed